CLINICAL TRIAL: NCT05061368
Title: The Effect of Oral Sildenafil on Exercise Capacity, Dyspnea and Cardiopulmonary Function in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Oral Sildenafil for Exercise Capacity, Dyspnea and Cardiopulmonary Function in COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00108944
Record Dates: First submitted 2021-08-16; First posted 2021-09-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Sildenafil; Pulmonary Vascular Function; Pulmonary Vascular Pressure; DLCO; Pulmonary Capillary Blood Volume; Dyspnea; Exercise Tolerance; Peak Oxygen Uptake; Cardiopulmonary Fitness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Double Blinded, Placebo Controlled Repeated Measures
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blinded: participants, investigators and outcome assessors are blinded to condition until data entry and analysis are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Experimental): Participants will be administered a 25 mg oral dose of sildenafil.
  Interventions: Drug: Sildenafil Citrate
- Placebo (Placebo Comparator): Participants will be administered an oral placebo indistinguishable from the sildenafil pill.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — Phosphodiesterase Type 5 inhibitor. Known to potentiate nitric oxide mediated vasodilation.
  Arms: Sildenafil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a condition characterized by airway obstruction. Patients with COPD experience significant shortness of breath on exertion. The mechanisms responsible for shortness of breath on exertion are well understood in moderate and severe COPD, but, are poorly understood in mild COPD where symptoms appear disproportionate to the degree of airway obstruction.

Mild COPD patients show an exaggerated breathing response to exercise, determined by the breathing response to carbon dioxide production (V̇E/V̇CO2). Recent work suggests that the increased V̇E/V̇CO2 during exercise in mild COPD is secondary to increased deadspace (i.e. lung regions with ventilation but no perfusion) and/or ventilation/perfusion (V̇A/Q) inequality (poor matching of ventilation to perfusion). Researchers have proposed that the increased deadspace or V̇A/Q inequality is secondary to pulmonary vascular dysfunction and hypoperfusion of the pulmonary capillaries.

Recently, we have shown that inhaled nitric oxide, a potent dilator of pulmonary vasculature, reduces shortness of breath and V̇E/V̇CO2, and improves exercise capacity in mild COPD. This preliminary finding suggests that pulmonary vascular dysfunction is an important contributor to exercise intolerance in mild COPD. Here, we aim to test whether sildenafil, an oral pulmonary vasodilator, can improve exercise tolerance and shortness of breath in mild COPD.

DETAILED DESCRIPTION:
COPD is a condition characterized by airway obstruction and is currently the 4th leading cause of death in Canada. Patients with COPD experience significant exertional dyspnea, which has been shown to reduce quality of life and physical activity, and increase risk of mortality. Much work has examined the mechanisms for dyspnea in moderate and severe COPD, but the mechanisms for dyspnea in patients with mild COPD, in whom symptoms are often disproportionate to the degree of airway obstruction, are not well understood. Mild COPD patients show an exaggerated ventilatory response to exercise, determined by the ventilatory response to carbon dioxide production (V̇E/V̇CO2), which is a key contributor to dyspnea and is predictive of mortality. Recent work suggests that the increased V̇E/V̇CO2 during exercise in mild COPD is secondary to increased deadspace (i.e. ventilation with no perfusion) and/or ventilation/perfusion (V̇ A/Q) inequality (i.e. poor matching of ventilation to perfusion). Researchers have proposed that the increased deadspace or V̇A/Q inequality is secondary to pulmonary vascular dysfunction and hypoperfusion of the pulmonary capillaries. Recently we have shown that iNO reduces dyspnea, and V̇E/V̇CO2, and improves exercise capacity in mild COPD, suggesting that pulmonary vascular dysfunction is an important contributor to exercise intolerance in mild COPD. Importantly, this work demonstrated that pulmonary NO mediated vasodilation pathways are intact, and are a viable target for improving exercise tolerance in mild COPD. Therefore, we hypothesize that sildenafil, which potentiates intrinsic NO mediated vasodilation mechanisms, will improve exercise tolerance in mild COPD.

Compared to disease free controls, mild COPD patients have a blunted diffusion capacity and pulmonary capillary blood volume response to exercise. In the supine position, which minimizes flow heterogeneity through removal of the coronal gravity-induced pressure gradient, diffusion capacity and pulmonary capillary blood volume responses to exercise were not corrected. The implication of this finding is that even mild COPD, there is a degree of permanent vascular destruction, in addition to reversible pulmonary vascular dysfunction. It is presently unknown when or if in the COPD severity continuum there is a transition from treatable pulmonary vascular dysfunction to irreversible pulmonary vascular destruction.

Sildenafil was previously tested in moderate to severe COPD with mixed success. Blanco et al. tested the effect of sildenafil (20 or 40 mg dose) on hemodynamics and gas exchange in a sample of patients with moderate to severe COPD. Eighty-five percent of the sample had pulmonary hypertension defined as mean pulmonary artery pressure >20 mmHg. Sildenafil significantly reduced pulmonary artery pressure at rest and during exercise (-6 and -11 mmHg respectively), and improved VA/Q inequality. Rietema et al. found no benefit of sildenafil (3x50mg daily for 3 months) on stroke volume (supine, rest/exercise) or exercise capacity in moderate to severe COPD. In a randomized, placebo controlled trial, sildenafil (3x20 mg daily, 3 months) did not improve pulmonary rehabilitation outcomes including cycle endurance time, 6 minute walk distance, or quality of life. It is not known why the promising reduction in pulmonary artery pressure and improved V̇A/Q matching did not translate to increased stroke volume or exercise capacity with chronic sildenafil dosing. Results may partially be explained by supine body positioning during measurement of stroke volume, and the generally late disease state of COPD patients. Pulmonary vascular dysfunction observed early in disease progression may transition to irrevocable vascular/pulmonary structural changes, for which iNO or sildenafil have limited utility. Accordingly, a secondary objective of the present study is to gain understanding of pathological vascular progression in COPD to identify the therapeutic window for pulmonary vascular intervention. We hypothesize that sildenafil will have greater cardiopulmonary benefit (increased diffusion capacity at rest and during exercise, greater decrease in pulmonary artery pressure) in early, mild COPD as compared to moderate-severe COPD, indicative of vascular dysfunction in mild COPD transitioning to vascular destruction in later disease states.

Trial Objectives

1. To examine the effect of acute oral sildenafil on maximal oxygen consumption (peak V̇O2) during exercise in the continuum of COPD
2. To examine whether acute oral sildenafil improves exertional dyspnea in COPD.
3. To examine the cardio-pulmonary effects and mechanisms of oral sildenafil.

Trial Design

Primary Study Endpoints/Secondary Endpoints Primary study endpoints for the proposed study are:

1. Exercise capacity as determined by maximal oxygen consumption (peak V̇O2).

   Secondary study endpoints for the proposed study are:
2. Dyspnea during exercise (modified Borg scale, 1-10)
3. Pulmonary function during exercise (V̇ E/V̇CO2, pulmonary capillary blood volume, diffusion capacity)
4. Cardiac output as determined by impedance cardiography.
5. Pulmonary artery pressure (estimated from rest/stress echocardiography).

Study Design

Randomized, double-blinded, placebo controlled cross-over design

Treatment: Sildenafil (oral), 25 mg; Placebo: Medical grade placebo pill

Seven sessions will be completed within an 8-week period in the following order:

Visit 1) Participant enrollment and familiarization, medical history, COPD assessment test (CAT), modified Medical Research Council (mMRC) dyspnea scale, standard pulmonary function test (PFT, including bronchodilator control) and a staged to maximal cardiopulmonary exercise test (CPET) with electrocardiography (ECG), pulse oximetry, and intermittent blood pressure and rating of perceived exertion (RPE, leg fatigue and dyspnea, modified Borg scale). A small blood sample will be collected via finger prick to measure hemoglobin (to correct DLCO). An additional venous blood sample will be collected for analysis of blood biomarkers to characterize participants including serum analysis of interleukin 6, c-reactive protein and tumor necrosis factor alpha.

Visits 2 and 3) Participants will be administered oral placebo/sildenafil (randomly ordered), wait for 30 minutes and then begin testing. Participants will undergo a staged to maximal CPET (gas exchange analysis, heart rate, cardiac output measured by impedance cardiography, blood pressure, RPE, arterial oxygen saturation).

Visits 4 and 5) Participants will be administered oral placebo/sildenafil (randomly ordered), wait for 30 minutes and then begin testing. Testing will start with measurement of resting diffusion capacity, pulmonary capillary blood volume (Vc), and membrane diffusion capacity (Dm) using the multiple fractional inspired oxygen (FIO2)-DLCO technique. Participants will then cycle at 40 W and 50% of peak work rate as determined from Visit 1, measurements will be repeated during steady-state exercise. Heart rate, oxygen saturation, and carboxyhemoglobin will be monitored throughout. A small blood sample will be collected via finger prick following each stage (rest, 40W, 50% of peak work rate) to measure hemoglobin to correct DLCO values.

Visit 6) Participants will undergo non-randomized control and then sildenafil rest and handgrip stress echocardiography. Echocardiography will be used to estimate cardiac volumes, function and pulmonary artery systolic pressure at rest and during handgrip stress. Isometric handgrip stress echocardiography was previously used in healthy and clinical populations to evoke marked cardiac stress without hyperpnoea- a major factor compromising image quality, particularly in COPD due to dynamic hyperinflation.

Visit 7) Participants will undergo chest computed tomography to characterize lung structure and emphysema.

Visit 1 is anticipated to take ~2 hours. Visits 2 and 3 are anticipated to take ~1.5 hours. Visits 4 and 5 are anticipated to take 2 hours. Visit 6 is anticipated to take 2 hours. Visit 7 is anticipated to take 1 hour. The anticipated total study duration is ~12 hours.

Data Analysis

A mixed-effects model will be used to evaluate the change in V̇O2peak with sildenafil. A two-way repeated measures ANOVA will be used to test for a difference in VO2peak response in mild COPD compared to COPD free controls. Two-way repeated measures ANOVA will be used to evaluate changes in dyspnea, cardiac output, ventilation, ventilatory efficiency (V̇E/V̇CO2), diffusion capacity and capillary blood volume during exercise. Variance in V̇O2peak changes will be explored using Pearson's regression and moderation analysis of echo-derived cardiac factors and pulmonary function/gas exchange. A three-way repeated measures ANOVA will be used to test for differences in pulmonary capillary blood volume response to sildenafil between mild and moderate COPD.

ELIGIBILITY:
Inclusion Criteria:

Participants will have COPD as defined as:

1. Post bronchodilator Forced Expiratory Volume in one second (FEV1) to Forced Vital Capacity (FVC) ratio (FEV1/FVC) below the lower limit of normal
2. FEV1 >30% of predicted (lower limit of GOLD severe COPD classification)

COPD Free Controls will have:

1. No diagnosis of COPD
2. Post bronchodilator Forced Expiratory Volume in one second (FEV1) to Forced Vital Capacity (FVC) ratio (FEV1/FVC) above the lower limit of normal
3. FEV1 >80% of predicted

Exclusion Criteria:

1. Absolute contraindication to exercise testing or an orthopedic condition that may limit exercise testing.
2. Pre-existing cardiac conditions (heart failure, congenital heart defect, valvular disease) that may limit exercise testing
3. A diagnosis of pulmonary hypertension preceding COPD
4. Current phosphodiesterase type-5 inhibitor, nitrate, opioid, azole antifungal, macrolide antibiotic, protease inhibitor, alpha blocker, riociguat, mifepristone or rifamycin use.
5. Pregnancy or lactation.
6. Women of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy throughout the study. Acceptable methods of contraception include tubal ligation, oral contraceptive, barrier methods (intra-uterine device, diaphragm, female condom, male condom). Abstinence is an acceptable form of contraception, only insofar as patients agree to use another acceptable method of birth control, preferably a barrier method, if they become sexually active.
7. Postmenopausal female participants must be amenorrheic for ≥12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | Within 20-25 minutes post-dose
  Maximal oxygen uptake (peak VO2)

SECONDARY OUTCOMES:
Dyspnea during exercise | Assessed every 2-minutes until completion of the exercise trial
  Modified Borg Scale (1-10)
Pulmonary function during exercise | Within 20-25 minutes post-dose
  VE/VCO2, pulmonary capillary blood volume, membrane diffusion capacity
Cardiac Output during exercise | Within 20-25 minutes post-dose
  Impedance Cardiography (l/min)
Pulmonary Artery Systolic Pressure | Assessed for five consecutive cardiac cycles and are measured in triplicate
  Estimated by tricuspid regurgitant jet velocity (echocardiography)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco I, Gimeno E, Munoz PA, Pizarro S, Gistau C, Rodriguez-Roisin R, Roca J, Barbera JA. Hemodynamic and gas exchange effects of sildenafil in patients with chronic obstructive pulmonary disease and pulmonary hypertension. Am J Respir Crit Care Med. 2010 Feb 1;181(3):270-8. doi: 10.1164/rccm.200907-0988OC. Epub 2009 Oct 29. PMID 19875684
- [Background] Phillips DB, Brotto AR, Ross BA, Bryan TL, Wong EYL, Meah VL, Fuhr DP, van Diepen S, Stickland MK; Canadian Respiratory Research Network. Inhaled nitric oxide improves ventilatory efficiency and exercise capacity in patients with mild COPD: A randomized-control cross-over trial. J Physiol. 2021 Mar;599(5):1665-1683. doi: 10.1113/JP280913. Epub 2021 Jan 25. PMID 33428233
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] Blanco I, Santos S, Gea J, Guell R, Torres F, Gimeno-Santos E, Rodriguez DA, Vilaro J, Gomez B, Roca J, Barbera JA. Sildenafil to improve respiratory rehabilitation outcomes in COPD: a controlled trial. Eur Respir J. 2013 Oct;42(4):982-92. doi: 10.1183/09031936.00176312. Epub 2013 Feb 21. PMID 23429918